CLINICAL TRIAL: NCT06476262
Title: Investigating Occupational Gaps After Mild Stroke: Prevalence, Explanatory Factors, and Impact on Quality of Life in a Single-Center Study
Brief Title: Occupational Gaps After Mild Stroke: a Single-Center Observational Study
Acronym: POPPAL
Status: Completed | Type: Observational
Sponsor: Grosmaire (Other)
Collaborators: Centre Hospitalier Sud Francilien (Other)
Responsible Party: Sponsor-Investigator, Grosmaire, OT, CRA, Clinique Les Trois Soleils
Organization: Clinique Les Trois Soleils (Other)
Other Study IDs: POPPAL
Record Dates: First submitted 2024-06-21; First posted 2024-06-26 (Actual); Last update posted 2024-06-26 (Actual); Status verified 2024-06

CONDITIONS: Stroke; Occupational Problems
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Behavioral: This research has only one arm. The intervention focuses on occupational issue — During the post-stroke consultation, each participant is invited to complete questionnaires on occupational gaps, mood disorders, fatigue, cognition, and quality of life.

SUMMARY:
The goal of this observational study is to investigate participation restrictions and their determinants in people after a mild stroke. The main questions it aims to answer are:

Do mRS score, time since stroke onset, cognitive disorders, mood disorders and fatigue negatively impact occupations after mild stroke?

Does an increased prevalence of occupational gaps correlate with a diminished quality of life following mild stroke?

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old,
* a diagnosis of stroke confirmed by cerebral imaging,
* an mRS score <3 at the post-stroke consultation,
* informed about the study
* not opposed to participation

Exclusion Criteria:

* cognitive dysfunction making participation in the study impossible,
* phasic disorders preventing comprehension of the questionnaires,
* neurological deficits prior to the stroke, a history of psychiatric disorders
* being under legal protection.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population was selected from the active file of stroke patients undergoing post-stroke consultation at the Centre Hospitalier Sud Francilien.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-02-13 (Actual); Primary Completion 2023-05-11 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Occupational Gaps Questionnaire | the OGQ was administred at the inclusion
  The Occupational Gaps Questionnaire (OGQ) assesses presence of occupational gaps in 28 activities, i.e. instrumental ADL, social- leisure- and work/work related activities. Two studies are published on occupational gaps. An occupational gap is defined as the gap that occurs between what an individual wants and needs to do and what he/she actually does.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression scale | HADS was asministred at the inclusion
  The Hospital Anxiety and Depression Scale (HADS) is a questionnaire widely used for detecting anxiety and depressive disorders.HADS comprises 14 items, seven of which relate to anxiety symptoms and seven to depressive symptoms. Each item is coded from 0 to 3. The scores for anxiety and depression can therefore vary from 0 to 21, depending on the presence and severity of the symptoms
Montreal Cognitive Assessment | MoCA was administred at the inclusion
  The Montreal Cognitive Assessment (MoCA) was designed as a rapid screening instrument for the detection of mild cognitive impairment. The MoCA assesses the following cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation.
Stroke Impact Scale | The SIS was administred at the inclusion
  The Stroke Impact Scale (SIS) is a stroke-specific, self-report, health status measure. It was designed to assess multidimensional stroke outcomes, including strength, hand function Activities of Daily Living / Instrumental Activities of Daily Living (ADL/IADL), mobility, communication, emotion, memory and thinking, and participation.
modified Ranking Scale | The mRS was administred at the inclusion
  The Modified Rankin Scale (MRS) is a single item, global outcomes rating scale for patients post-stroke. It is used to categorize level of functional independence with reference to pre-stroke activities rather than on observed performance of a specific task.
Fatigue Severity Scale | The FSS was administred at the inclusion
  The Fatigue Severity Scale (FSS) is a 9-item scale which measures the severity of fatigue and its effect on a person's activities and lifestyle in patients with a variety of disorders.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe T Duret, MD, Principal Investigator — Clinique Les Trois Soleils
Locations (1):
- Clinique Les Trois Soleils, Boissise-le-Roi, France

IPD SHARING:
Plan to Share IPD: No